CLINICAL TRIAL: NCT00408603
Title: A Phase 2 Open-Label, Multicenter Study of SNS-595 Injection in Patients With Platinum-Resistant Ovarian Cancer
Brief Title: Safety and Efficacy Clinical Study of SNS-595 in Patients With Platinum-Resistant Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0010
Record Dates: First submitted 2006-12-05; First posted 2006-12-07 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Epithelial Ovarian Cancer
Keywords: second line treatment; platinum resistant; ovary; ovaries; cancer; epithelial; carcinomas; tumor
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Neoplasms; Carcinoma | interventions — vosaroxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All study patients (Experimental): All patients will receive voreloxin injection
  Interventions: Drug: Voreloxin Injection

INTERVENTIONS:
Drug: Voreloxin Injection — All patients in initial dose level receive voreloxin injection at 48 mg/m2 administered once every 21 days up to 6 cycles. Subsequent levels are of 60 mg/m2 or 75 mg/m2 every 28 days up to 6 cycles if safety acceptable.
  Other Names: SNS-595, vosaroxin, Qinprezo

SUMMARY:
The purpose of this study is to evaluate the objective response rate, safety and identify potential biomarkers in platinum-resistant ovarian cancer patients treated with voreloxin injection given on a 28-day cycle.

DETAILED DESCRIPTION:
Other objectives of this study are to evaluate Progression-free survival and measure CA-125 response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented epithelial ovarian cancer, primary peritoneal carcinoma, or fallopian tube cancer
* Completed at least one Platinum Based Therapy (PBT) regimen (carboplatin, cisplatin, or another organoplatinum compound).
* Evidence of platinum-resistant disease, relapse/progression within 6 months of the completion of PBT, or intolerant to PBT (inability to receive PBT due to hypersensitivity reactions to platinum)
* Patients with primary platinum-resistant disease are allowed to receive no more than one nonplatinum cytotoxic regimen and no more than one noncytotoxic regimen for the management of recurrent or persistent disease after the development of primary platinum-resistance.
* Measurable disease per GOG-RECIST criteria
* GOG Performance Status of 0 or 1

Exclusion Criteria:

* Radiotherapy, chemotherapy, and hormonal, cytokine, or targeted therapy, within 3 weeks (nitrosurea or mitomycin C within 6 weeks) prior to the anticipated first day of treatment.
* Monoclonal antibody therapy within 4 weeks prior to clinical study entry
* Unresolved or impending bowel obstruction
* Other active malignancies or other malignancies within the last 12 months except nonmelanoma skin cancer or cervical intraepithelial neoplasia
* Prior radiotherapy to more than 25% of the marrow space
* Requiring hemodialysis or peritoneal dialysis
* Myocardial infarction or cerebrovascular accident/transient ischemic attack within the 6 months prior to the anticipated first day of treatment
* Thromboembolic event (deep vein thrombosis [DVT] or pulmonary embolus [PE]) within 28 days prior to the anticipated first day of treatment
* History of active CNS metastases
* Any other medical, psychological, or social condition that would contraindicate the patient's participation in the clinical study due to safety or compliance with clinical study procedures.

Please note: There are additional inclusion/exclusion criteria for this study. Please contact the study center for additional information and to determine if you meet all study criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 183 (Actual)
Dates: Start 2006-12-20 (Actual); Primary Completion 2010-06-09 (Actual); Study Completion 2010-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunesis Medical Monitor, MD, Study Director — Sunesis Pharmaceuticals
Locations (20):
- United States (14):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Gynecologic Oncology Associates, Newport Beach, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Stanford University, Stanford, California
  - Medstar Research Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Oncology Specialists, S.C. at Luthern General Advanced Care Center, Park Ridge, Illinois
  - Louisville Oncology Clinical Research Program, Louisville, Kentucky
  - The Harry and Jeanette Weinberg Institute at Franklin Square, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - Kaiser Permanente NW Region, Portland, Oregon
  - University of Pittsburgh Medical Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Hall and Martin, MD's, P.C., Knoxville, Tennessee
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency at Centre for Southern Interior, Kelowna, British Columbia
  - BC Cancer Agency at Fraser Valley Centre, Surrey, British Columbia
  - BC Cancer Agency at Vancouver, Vancouver, British Columbia
  - BC Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - Juravinski Cancer Centre Department of Oncology, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of individual participants experiencing Serious Adverse Events, post trial completion

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 48 mg/m2: All Stage 1 patients will receive voreloxin injection
  Voreloxin Injection: All Stage 1 patients in initial dose level receive voreloxin injection at 48 mg/m2 administered once every 21 days up to 6 cycles.
- Stage 60 mg/m2: Following safety of 48 mg/m2 group, next Stagel is 60mg/m2 at 28 day periods up to 6 cycles.
- Stage 75 mg/m2: Following safety of 60 mg/m2 group, next Stage is 75 mg/m2 at 28 day periods up to 6 cycles.
Period: Overall Study
Arm/Group | Stage 48 mg/m2 | Stage 60 mg/m2 | Stage 75 mg/m2
Started | 69 | 39 | 75
Completed | 65 | 37 | 35
Not Completed | 4 | 2 | 40

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- 48 mg/m2: 48 mg/m2 every 21 days
- 60 mg/m2: 60 mg/m2 every 28 days
- 75 mg/m2: 75 mg/m2 every 28 days
- Total: Total of all reporting groups
Arm/Group | 48 mg/m2 | 60 mg/m2 | 75 mg/m2 | Total
Number analyzed (Participants) | 65 | 37 | 35 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9.87) | 62.7 (10.51) | 57.6 (12.13) | 60.1 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 37 | 35 | 137
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 65 | 37 | 35 | 137
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5 | 1 | 2 | 8
  Black or African | 4 | 1 | 1 | 6
  White or Caucasian | 56 | 35 | 31 | 122
  Other, Philippines | 0 | 0 | 1 | 1
Height (cm) [Mean (Standard Deviation); unit: cm] | 162.4 (6.75) | 161.9 (7.01) | 163.9 (7.01) | 162.7 (6.88)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 75.1 (17.21) | 71.2 (20.52) | 69.9 (15.39) | 72.7 (17.76)
BSA (m2) [Mean (Standard Deviation); unit: m2] | 1.8 (0.2) | 1.7 (0.24) | 1.8 (0.2) | 1.8 (0.21)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (CR+PR) Per Investigator Assessment Based on GOG-RECIST Criteria
Description: Response rate was calculated per investigator's tumor assessment based on GOG-RECIST, which includes radiographic imaging, physical examination results, and CA-125 levels. No independent review of CT scans (lesion assessments) was performed. CR: disappearance of all target and nontarget lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Normalization of CA125, if elevated at baseline, is required for ovarian carcinoma studies. PR is >= 30% decrease in the sum of LD of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of nontarget lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required.
Time Frame: GOG-RECIST assessment obtained on cycle2, 4 and 6 Day 21for patients treated with 48 mg/m2 SNS-595 and Day 28 for patients treated with 60 mg/m2, through 28 (±14) days afte the last treatment at the end of safety follow up period
Population: Safety Population which included all patients who received any amount of vosaroxin
Measure: Count of Participants; unit: Participants
Groups:
- Total: Overall
Arm/Group | 48 mg/m2 | 60 mg/m2 | 75 mg/m2 | Total
Number analyzed (Participants) | 65 | 37 | 35 | 137
Participants | 7 | 4 | 3 | 14

2. Secondary Outcome: Progression-free Survival (PFS) Using Kaplan-Meier Methods
Description: PFS is the the time between the date the patient first received Vosaroxin and the earliest date of disease progression.
  For patients who experienced disease progression, the date of disease progression will be the earliest date on which disease progression is indicated based on the rules.
  For patients who died with no indication of disease progression, the date of death will be the earliest date on which death is documented based on the rules.
  For patients who have no indication of disease progression or death, the censoring date will be the Date of Confirmed Contact from the last Survival Follow-Up CRF, or if not in survival follow-up, then the Assessment Date from the last GOG-RECIST CRF, or if no response assessment available, Date of Last Visit / Contact from Extended Treatment Completion CRF if in extended treatment, or from Cycle 6 Completion / Early Termination CRF if not in extended treatment.
Time Frame: From the first teratment of Vosaroxin to the end of Cycle 6 or 28 days after the last treatment at the end of safety follow up period if continued in the extended treatment period
Population: Safety population which included all patients who received any amount of vosaroxin
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | 48 mg/m2 | 60 mg/m2 | 75 mg/m2 | Total
Number analyzed (Participants) | 65 | 37 | 35 | 137
Days | 83 [49 to 90] | 61 [53 to 134] | 103 [53 to 167] | 81 [57 to 93]

ADVERSE EVENTS:
Time Frame: Approximately 50% of patients were assessed for AEs for 112 days or less and the other approximate 50% were assessed for 112 to 700 days.
Arm/Group | 48 mg/m2 | 60 mg/m2 | 75 mg/m2 | Total
All-Cause Mortality (participants affected / at risk) | 7/65 | 2/37 | 3/35 | 11/137
Serious Adverse Events (participants affected / at risk) | 15/65 | 9/37 | 14/35 | 38/137
Other Adverse Events (participants affected / at risk) | 63/65 | 37/37 | 35/35 | 135/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 48 mg/m2 (N=65) | 60 mg/m2 (N=37) | 75 mg/m2 (N=35) | Total (N=137)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 10 | 15
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 4
Fatigue (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 0 | 3
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0 | 0 | 1
Bacillus infection (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 1
Catheter bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Brain stem syndrome (Nervous system disorders) | 0 | 0 | 1 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 48 mg/m2 (N=65) | 60 mg/m2 (N=37) | 75 mg/m2 (N=35) | Total (N=137)
Anaemia (Blood and lymphatic system disorders) | 14 | 14 | 13 | 41
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 1 | 7
Leukopenia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 8
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 21 | 8 | 18 | 47
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 2 | 2 | 5
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 0 | 4
Blepharospasm (Eye disorders) | 0 | 0 | 1 | 1
Dark circles under eyes (Eye disorders) | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 2 | 3
Lacrimation increased (Eye disorders) | 1 | 1 | 0 | 2
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 1 | 1
Photopsia (Eye disorders) | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 3 | 1 | 2 | 6
Visual disturbance (Eye disorders) | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 16 | 9 | 9 | 34
Abdominal hernia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Abdominal mass (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 22 | 7 | 12 | 41
Abdominal pain lower (Gastrointestinal disorders) | 2 | 2 | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 5 | 2 | 1 | 8
Abdominal tenderness (Gastrointestinal disorders) | 3 | 0 | 3 | 6
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 5 | 1 | 3 | 9
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 25 | 23 | 11 | 59
Diarrhoea (Gastrointestinal disorders) | 26 | 12 | 17 | 55
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 3 | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 19 | 4 | 5 | 28
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 6 | 1 | 1 | 8
Gastric hypomotility (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 5 | 6 | 1 | 12
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3 | 1 | 4
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 51 | 27 | 24 | 102
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Salivary gland disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 3 | 1 | 6
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 19 | 8 | 3 | 30
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Tongue oedema (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 26 | 19 | 17 | 62
Asthenia (General disorders) | 2 | 1 | 2 | 5
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 2
Chills (General disorders) | 8 | 1 | 4 | 13
Early satiety (General disorders) | 1 | 2 | 1 | 4
Face oedema (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 52 | 30 | 27 | 109
Gait disturbance (General disorders) | 0 | 1 | 1 | 2
Hernia pain (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 4 | 0 | 0 | 4
Infusion site bruising (General disorders) | 2 | 0 | 0 | 2
Infusion site erythema (General disorders) | 1 | 0 | 0 | 1
Infusion site rash (General disorders) | 1 | 0 | 0 | 1
Infusion site reaction (General disorders) | 1 | 0 | 1 | 2
Injection site erythema (General disorders) | 0 | 1 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 2 | 2
Irritability (General disorders) | 1 | 0 | 0 | 1
Local swelling (General disorders) | 0 | 1 | 0 | 1
Nodule (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 1 | 1 | 5
Oedema (General disorders) | 3 | 2 | 1 | 6
Oedema peripheral (General disorders) | 8 | 6 | 2 | 16
Pain (General disorders) | 3 | 2 | 6 | 11
Peripheral coldness (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 12 | 3 | 8 | 23
Temperature intolerance (General disorders) | 0 | 0 | 3 | 3
Visceral oedema (General disorders) | 1 | 1 | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 2 | 3
Abdominal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 2
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 3 | 0 | 0 | 3
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 3 | 0 | 1 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 5 | 2 | 0 | 7
Neutropenic infection (Infections and infestations) | 1 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 1 | 2 | 4
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 2
Perianal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 2
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 5
Urinary tract infection (Infections and infestations) | 4 | 5 | 10 | 19
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 1
Vaginal candidiasis (Infections and infestations) | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 1
Breath sounds abnormal (Investigations) | 1 | 2 | 1 | 4
Haemoglobin decreased (Investigations) | 1 | 1 | 1 | 3
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 1
Lymph node palpable (Investigations) | 0 | 1 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 6 | 6 | 3 | 15
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 2
White blood cell count increased (Investigations) | 0 | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 27 | 15 | 12 | 54
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 5 | 2 | 6 | 13
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 7 | 6 | 18
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5 | 3 | 11
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 3 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | 7 | 26
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 4
Jaw disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 2 | 10
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Spinal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 12 | 2 | 5 | 19
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 17 | 4 | 6 | 27
Headache (Nervous system disorders) | 15 | 5 | 4 | 24
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 2
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 2
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 1
Neuropathy (Nervous system disorders) | 2 | 1 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 1 | 2 | 5
Pallanaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 2 | 4
Parosmia (Nervous system disorders) | 2 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 2 | 3
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1 | 2
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 3 | 6
Confusional state (Psychiatric disorders) | 2 | 0 | 2 | 4
Depression (Psychiatric disorders) | 8 | 1 | 3 | 12
Insomnia (Psychiatric disorders) | 3 | 8 | 2 | 13
Bladder discomfort (Renal and urinary disorders) | 1 | 0 | 1 | 2
Bladder pain (Renal and urinary disorders) | 1 | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 2 | 2 | 6
Haematuria (Renal and urinary disorders) | 4 | 0 | 1 | 5
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 2
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 2 | 2 | 4
Pollakiuria (Renal and urinary disorders) | 2 | 3 | 3 | 8
Proteinuria (Renal and urinary disorders) | 3 | 0 | 0 | 3
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 2 | 0 | 1 | 3
Genital pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 2
Vaginal discharge (Reproductive system and breast disorders) | 2 | 0 | 0 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 0 | 1 | 5
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 7 | 24
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 6 | 7 | 33
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 5
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 9 | 22
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 40 | 24 | 26 | 90
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 6
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 6
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 2 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 9
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Skin nodule (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 2
Flushing (Vascular disorders) | 2 | 2 | 3 | 7
Hot flush (Vascular disorders) | 6 | 1 | 5 | 12
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 2 | 4
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
No statistical testings were performed to compare any of the treatment groups. No p-values or odds ratios were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days